CLINICAL TRIAL: NCT03043716
Title: Long-term Observation of Adherence and Efficacy of Patients With a Positive Airway Pressure (PAP) Therapy With Use of Telemonitoring
Brief Title: Long-term Observation of PAP-therapy With Telemonitoring: Telemedicine Registry TelePAP
Acronym: TelePAP
Status: Active, not recruiting | Type: Observational
Sponsor: ResMed (Industry)
Collaborators: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: TelePAP_Protokoll_V02_17072017
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea; Central Sleep Apnea; Mixed Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PAP therapy with telemonitoring — Patients will receive a prescription for PAP therapy in the course of their clinical Routine pathway and afterwards be asked to enrol in the registry. The will be asked if they are willing to use telemonitoring technology.

SUMMARY:
Telemonitoring for Positive Airway Pressure (PAP) therapy might help to establish and maintain long-term therapy adherence and thus support the beneficial effects of PAP therapy on long-term outcomes.

DETAILED DESCRIPTION:
Airway obstructions, airflow resistance by partial occlusion of the airways or central sleep-breathing disorders, where the respiratory effort is reduced or stops, cause a reduction in airflow and lead to arousals from sleep and disturbances in gas exchange during sleep. The negative consequences manifest in increases of blood pressure, higher workload for the heart and daytime sleepiness. PAP (positive airway pressure) treats sleep-related breathing disorders. It applies pressure to nose and mouth to keep the airway from collapsing and provides pressure support to assist the respiratory muscles. The efficacy of the therapy is measured with apnoea- and hypopnoea-indices that count the total number of apnoeic events at night. To ensure an efficacious and efficient therapy, pressures have to be adjusted correctly and the patient needs to use PAP regularly.

Telemonitoring is information and communication technology to exchange sleep data and to provide clinical guidance over distances. There is no defined spectrum of technology. It can comprise phone calls, video support or interaction programs via the internet. Some studies point to advantages of telemonitoring in keeping compliance upright, increase usage hours and some also point to economic advantages. However, we do not have conclusive data from large trials with telemonitoring on the long-term that would show conclusive effects, be it from the side of a patient or from a cost and labour perspective of providers or the healthcare sector. Still, there are uncertainties regarding data safety, reimbursement or connectivity of different systems.

No long-term data of PAP therapy under telemonitoring and its effect on compliance and therapy outcomes is available by now.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* New indication for a prescription of a Telemonitoring (AirViewTM)-capable ResMed PAP-device
* Consent to use the telemonitoring System AirViewTM (ResMed GmbH & Co KG)
* Signed Informed Consent

Exclusion Criteria:

- Pregnant and breastfeeding persons

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult individuals with an indication for a therapy with positive airway pressure. Sleep breathing disorders can be obstructive (obstructive sleep apnea, OSA) or central (CSA) ranging from mild forms (apnoea-hypopnoea-index ˃ 5 and ˂ 15) over moderate (AHI ˃15 and ˂30) or severe (AHI ˃ 30).
Sampling Method: Non-Probability Sample
Enrollment: 14147 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Usage Patterns of PAP therapy with telemonitoring, assessed by data continuously recorded by the device and transferred via telemonitoring | 24 months
  Usage Patterns are hours/night and nights/month that therapy has been used. Telemonitoring enables the physician to remotely supervise device usage. Usage will be assessed through data recordings of the device: Days of usage >3hours; Days of usage <3 hours; total recorded days; mean daily usage (minutes); total usage hours (h)

SECONDARY OUTCOMES:
Sleep disorders, assessed by personally questioning the Patient at baseline and at 24 months follow-up | 24 months
  Sleep disorders are snoring, insomnia, hypersomnia, depression, restless legs syndrome as assessed by anamnesis.
Therapy efficacy, assessed through changes in AHI and HI comparing baseline with 24 months follow-up | 24 months
  Efficacy is measured through changes in Apnea-Hypopnea-Index AHI (numbers of apneas - reduction of airflow by >90% for at least 10 seconds - and hypopneas - reduction of airflow by >30% for at least 10 seconds with a 4% decrease of Oxygen Saturation - divided by hours of sleep), AI - apnea index (apneas per hour), HI hypopnea index (hypopneas per hour).
Quality of Life, assessed with the Functional Outcomes of Sleep Questionnaire (FOSQ) comparing the score at baseline with the 24 months follow-up | 24 months
  The Functional Outcomes of Sleep Questionnaire had been developed to comprehensively capture the impact of sleeping disorders in relevant daily activities as for instance general activity, vigilance, intimacy, fitness and social life.
Factors leading to therapy Termination, assessed by personally questioning a Patient or Consulting a physician at time of follow-up | 24 months
  Possible causes for therapy Termination are assessed: Lost-to-follow-up, no interest in therapy, changed physician, no therapy benefits, Hospital stay, death

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Grüger, Dr, Principal Investigator — Grand Arc Düsseldorf
Locations (6):
- Germany (6):
  - Schlaf- und Beatmungszentrum Blaubeuren, Blaubeuren Abbey, Baden-Wurttemberg
  - Ambulante Schlafmedizin Herold/Kaa, Fürth, Bavaria
  - Klinikum Nürnberg-Med Klinik 3, Nuremberg, Bavaria
  - Klinik für Schlafmedizin Düsseldorf Grand Arc, Düsseldorf, North Rhine-Westphalia
  - Ruhrlandklinik Essen, Essen, North Rhine-Westphalia
  - Zentrum für Schlafmedizin Dr. Warmuth, Berlin